CLINICAL TRIAL: NCT02630485
Title: Graceful Lifestyle Changes Intervention Study for Women With PCOS and Infertility
Brief Title: Graceful Lifestyle Changes Study for PCOS and Infertility
Acronym: GLC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: H13-02964
Record Dates: First submitted 2015-11-30; First posted 2015-12-15 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Polycystic Ovary Syndrome; Infertility
Keywords: Randomized Controlled Trial
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility | interventions — Inositol; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Graceful Lifestyle Changes & MYO (Experimental): The 12-week lifestyle intervention will incorporate three lifestyle changes: a low-glycemic diet, increased exercise, and stress reduction through meditation and mindfulness.
  In addition, this group will take myo-inositol (6 grams in juice or water every morning).
  Interventions: Behavioral: Graceful Lifestyle Changes; Dietary Supplement: Myo-inositol
- Graceful Lifestyle Changes (Experimental): The 12-week lifestyle intervention will incorporate three lifestyle changes: a low-glycemic diet, increased exercise, and stress reduction through meditation and mindfulness.
  In addition, this group will take a white powder placebo (6 grams in juice or water every morning).
  Interventions: Behavioral: Graceful Lifestyle Changes
- Letrozole & MYO (Placebo Comparator): The women assigned to the fertility medication group will be prescribed letrozole. The initial dose will be 5 mg daily for five days and the dose can be increased by 2.5 mg to a total daily dose of 7.5 mg if necessary depending on ovulatory response, as in clinical practice. This treatment regimen will continue for three cycles (approximately the same period of time as the treatment group) or until pregnancy is achieved.
  In addition, this group will take myo-inositol (6 grams in juice or water every morning).
  Interventions: Dietary Supplement: Myo-inositol; Drug: Letrozole
- Letrozole (Placebo Comparator): The women assigned to the fertility medication group will be prescribed letrozole. The initial dose will be 5 mg daily for five days and the dose can be increased by 2.5 mg to a total daily dose of 7.5 mg if necessary depending on ovulatory response, as in clinical practice. This treatment regimen will continue for three cycles (approximately the same period of time as the treatment group) or until pregnancy is achieved.
  In addition, this group will take a white powder placebo (6 grams in juice or water every morning).
  Interventions: Drug: Letrozole

INTERVENTIONS:
Behavioral: Graceful Lifestyle Changes — Participants will be educated in small groups of 8-10. A wellness booklet designed by physicians and researchers at Grace Fertility Centre will be provided.The target diet for our study is 45% carbohydrates and 55 grams of glycemic load. Participants will keep a 3-day food diary at baseline, 4, 8 and 12 weeks. Secondly, participants will be provided a pedometer and a goal to reach 10,000 steps a day. The third aspect of the program will be to decrease overall stress through mindfulness. Educational sessions will be held to teach the relaxation response and meditation techniques such as breathing and grounding exercises. Participants will be required to meditate for at least 20 minutes each day and record this.
  Other Names: GLC
  Arms: Graceful Lifestyle Changes; Graceful Lifestyle Changes & MYO
Dietary Supplement: Myo-inositol — Myo-inositol will be consumed in juice or water every morning (6 grams) for 12 weeks.
  Other Names: Inositol; MYO
  Arms: Graceful Lifestyle Changes & MYO; Letrozole & MYO
Drug: Letrozole — Letrozole will be administered to patients. The initial dose will be 5 mg daily for five days and the dose can be increased by 2.5 mg to a total daily dose of 7.5 mg if necessary depending on ovulatory response, as in clinical practice. This treatment regimen will continue for three cycles (approximately the same period of time as the treatment group) or until pregnancy is achieved.
  Arms: Letrozole; Letrozole & MYO

SUMMARY:
The purpose of this study is to help women with PCOS to improve their symptoms and ovulation rate through a lifestyle intervention program which introduces a specific diet, a physical activity regimen and mindfulness exercises to improve psychological well-being and overall health.

DETAILED DESCRIPTION:
1) Purpose

The purpose of this study is to:

1. assess if implementing lifestyle changes through instruction and coaching is as effective as standard ovulation-induction therapy,
2. evaluate if myo-inositol is an effective addition to both lifestyle intervention and standard fertility medications, and
3. evaluate how each of four main sub-types of PCOS will respond to our lifestyle intervention program.

2) Hypothesis:

The investigators hypothesize that implementing lifestyle changes in women with PCOS will help restore ovulation by balancing reproductive hormones and increasing sensitivity to insulin. Lifestyle changes will also help to manage common PCOS symptoms and therefore, increase psychological well-being and quality of life in this population of women. In addition to a low-glycemic diet, physical activity, and stress reduction, a diet supplemented with myo-inositol will create further hormonal homeostasis and improve metabolic functioning. Finally, the investigators believe that the distinct sub-types of PCOS will respond differently to the proposed lifestyle intervention program and therefore, this will demonstrate that diet, activity and stress reduction is an effective approach to fertility for some individuals, but not others.

3) Justification:

Polycystic ovary syndrome (PCOS) is a heterogenous condition characterized by chronic anovulation and increased androgens (either as clinical or biochemical manifestations) according to the original NIH criteria. Since then, polycystic ovaries on ultrasound assessment has been included as an additional feature in the Rotterdam criteria and a diagnosis is made if a woman has any two of these three features. Very little information is known about why PCOS can present differently among individuals and which lifestyle factors are the cause or the effect. Many women with PCOS have difficulty conceiving due to infrequent ovulation. Evidence suggest that diet, activity and stress levels influence ovulation and affect the response of the ovaries to fertility medications or pregnancy success to fertility treatments.

To this date, there have been no studies conducted incorporating diet, exercise, and stress reduction in a cohesive intervention program for women with PCOS trying to conceive. Recent studies have suggested that women with PCOS can significantly benefit from specific lifestyle changes such as eating a low glycemic diet, increasing activity level, and reducing stress however, these studies have had several limitations such as high-drop out rates, lack of PCOS phenotypes included, and small cohort sizes. Also, most studies have focused on only one major lifestyle change, such as diet, which is not as powerful as combining diet, exercise and stress reduction. Finally, mindfulness and meditation as a means to decrease stress has yet to be studied in a PCOS cohort. The relaxation response is a powerful tool that has been proven to be effective in stress-related diseases such as cancer, cardiovascular disease and mental disorders. Since women with PCOS tend to have high levels of stress, inducing the relaxation response through mindfulness may be an effective treatment for this cohort.

4) Objectives

1. To determine if lifestyle changes are effective at restoring ovulation without the use of a commonly used fertility treatment.
2. To determine if myo-inositol improves the restoration of ovulation and insulin resistance in women with polycystic ovary syndrome (PCOS).
3. To evaluate how each of four main sub-types of PCOS will respond to our lifestyle intervention program.

5) Research Method:

Women with PCOS will be randomly assigned to one of two groups: the GLC group, which will participate in our "Graceful Lifestyle Changes" program and an oral fertility medication group, which will be prescribed letrozole. Within each of these two groups, participants will be further divided randomly to consume either myo-inositol or a placebo.

The GLC group will meet with physicians and educators, in small groups of 8-10 participants, once a week for 12 weeks. Each week will consist of an educational portion which will coach women on how to consume a low-glycemic diet, the benefits of walking 10,000 steps a day, and how to induce the relaxation response to decrease stress. A wellness booklet designed and provided by clinicians at Grace Fertility Centre will outline the main ideas being taught. Participants in the GLC group will be required to record their daily food intake to maintain a daily target of 45% carbohydrates and 55 grams of glycemic load a daily, which is similar to previous low-glycemic diet intervention studies. Lists will be provided outlining foods that are either low, medium, or high in glycemic load. Participants will be advised to eat as many low glycemic foods as possible and to limit the high glycemic load foods. They will also be provided with a pedometer to measure the number of steps being walked each day. Lastly, these participants will practice relaxation response exercises for twenty minutes each day and will record which exercises they performed in their daily diary.

Participants will complete a 3-day diet diary report as well as a physical activity report based on their pedometer recordings during the baseline, 4th, 8th, and 12th weeks. Participants will also receive a phone call from a trained researcher to complete a 24-hour diet recall at the end of the 2nd, 6th, and 10th weeks. This recall will assess all food consumed in the previous 24 hours. These combined methods will aim to:

* assess overall compliance to the low-glycemic diet
* provide information on the length of time participants take to comply
* evaluate any fluctuations in eating habits
* compare two types of nutritional assessment to each other

Compliance to the physical activity portion will be measured through daily pedometer recordings made by the participant. Compliance to the meditation and relaxation exercises will be measured by daily reports. Compliance will be ensured additionally through weekly check-ins/weigh-ins, weekly education sessions, and frequent email reminders with tips and motivators to stay on track.

The use of clomiphene citrate to treat anovulatory infertility is common. However, in agreement with what the investigators have observed in clinical practice, recent evidence has suggested that letrozole is more effective than clomiphene citrate in achieving ovulation. Additionally, letrozole may be more beneficial since it does not negatively affect the endometrial thickness. However, up to 40% of women may not ovulate with oral fertility treatments alone. Newer evidence suggests that diet, activity and stress levels influence ovulation and affect the response of the ovaries to fertility treatments.

ELIGIBILITY:
Inclusion Criteria:

* all women with PCOS trying to conceive who are between 18 and 37 years of age (PCOS will be defined using the Rotterdam criteria)

Exclusion Criteria:

* women who have already began fertility treatment
* women who are taking myo-inositol or have taken it in the past three months
* women being treated for or who have a history of an eating disorder

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-03 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Ovulation Occurence | 12 weeks
  Ovulation is the primary outcome and expressed as any ovulation (categorical "yes" or "no") during the 12-week (84-day) study. This length allows observation of 3 potential ovulatory cycles. The upper limit of a normal ovulatory cycle is 35 days, so to accommodate for this, documentation of ovulation with a progesterone test may extend to the end of week 14.
Ovulation Frequency | 12 weeks
  Ovulation is the primary outcome can be expressed in according to frequency (nominal "0", "1", "2, or "3") during the 12-week (84-day) study. This length allows observation of 3 potential ovulatory cycles. The upper limit of a normal ovulatory cycle is 35 days, so to accommodate for this, documentation of ovulation with a progesterone test may extend to the end of week 14.

SECONDARY OUTCOMES:
Conception | 12 weeks
  If ovulation occurs but menses does not follow, a pregnancy test will be administered.
Stress | 12 weeks
  Stress will be assessed by the Depression Anxiety and Stress Scale (DASS) at the beginning and end of the 12 weeks.
Anxiety | 12 weeks
  Anxiety will be assessed by the Depression Anxiety and Stress Scale (DASS) at the beginning and end of the 12 weeks.
Depression | 12 weeks
  Depression will be assessed by the Depression Anxiety and Stress Scale (DASS) at the beginning and end of the 12 weeks.
Quality of Life | 12 weeks
  Quality of life will be assessed by the Fertility Quality of Life Questionnaire (FertiQoL) at the beginning and end of the 12 weeks..

CONTACTS AND LOCATIONS:
Overall Officials: Anthony P Cheung, MBBS MPH MBA, Principal Investigator — Grace Fertility Centre & Reproductive Medicine

REFERENCES:
- [Background] Barr S, Reeves S, Sharp K, Jeanes YM. An isocaloric low glycemic index diet improves insulin sensitivity in women with polycystic ovary syndrome. J Acad Nutr Diet. 2013 Nov;113(11):1523-1531. doi: 10.1016/j.jand.2013.06.347. Epub 2013 Aug 30. PMID 23999280
- [Background] Barnard L, Ferriday D, Guenther N, Strauss B, Balen AH, Dye L. Quality of life and psychological well being in polycystic ovary syndrome. Hum Reprod. 2007 Aug;22(8):2279-86. doi: 10.1093/humrep/dem108. Epub 2007 May 30. PMID 17537782
- [Background] Costantino D, Minozzi G, Minozzi E, Guaraldi C. Metabolic and hormonal effects of myo-inositol in women with polycystic ovary syndrome: a double-blind trial. Eur Rev Med Pharmacol Sci. 2009 Mar-Apr;13(2):105-10. PMID 19499845
- [Background] Dunaif A. Insulin resistance and the polycystic ovary syndrome: mechanism and implications for pathogenesis. Endocr Rev. 1997 Dec;18(6):774-800. doi: 10.1210/edrv.18.6.0318. PMID 9408743
- [Background] Hutchison SK, Stepto NK, Harrison CL, Moran LJ, Strauss BJ, Teede HJ. Effects of exercise on insulin resistance and body composition in overweight and obese women with and without polycystic ovary syndrome. J Clin Endocrinol Metab. 2011 Jan;96(1):E48-56. doi: 10.1210/jc.2010-0828. Epub 2010 Oct 6. PMID 20926534
- [Background] Ludwig DS, Kabat-Zinn J. Mindfulness in medicine. JAMA. 2008 Sep 17;300(11):1350-2. doi: 10.1001/jama.300.11.1350. No abstract available. PMID 18799450
- [Background] Matchim Y, Armer JM, Stewart BR. Effects of mindfulness-based stress reduction (MBSR) on health among breast cancer survivors. West J Nurs Res. 2011 Dec;33(8):996-1016. doi: 10.1177/0193945910385363. Epub 2010 Oct 18. PMID 20956583
- [Background] Papaleo E, Unfer V, Baillargeon JP, De Santis L, Fusi F, Brigante C, Marelli G, Cino I, Redaelli A, Ferrari A. Myo-inositol in patients with polycystic ovary syndrome: a novel method for ovulation induction. Gynecol Endocrinol. 2007 Dec;23(12):700-3. doi: 10.1080/09513590701672405. Epub 2007 Oct 10. PMID 17952759
- [Background] Unfer V, Carlomagno G, Dante G, Facchinetti F. Effects of myo-inositol in women with PCOS: a systematic review of randomized controlled trials. Gynecol Endocrinol. 2012 Jul;28(7):509-15. doi: 10.3109/09513590.2011.650660. Epub 2012 Feb 1. PMID 22296306
- [Derived] Cutler DA, Shaw AK, Pride SM, Bedaiwy MA, Cheung AP. A randomized controlled trial comparing lifestyle intervention to letrozole for ovulation in women with polycystic ovary syndrome: a study protocol. Trials. 2018 Nov 16;19(1):632. doi: 10.1186/s13063-018-3009-5. PMID 30445999